CLINICAL TRIAL: NCT01047722
Title: Bleeding Volume Test: A Double-Blind Crossover Randomized Clinical Trial of an In-Vivo On-Line Test for Aspirin Effect and Resistance
Brief Title: In-Vivo Bleeding Volume Test for Platelet-Aspirin Interaction
Acronym: Aspirin-BVT
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Klein, Jeffrey A., M.D. (Individual)
Responsible Party: Principal Investigator, Jeffrey Alan Klein, MD, Principal Investigator, Klein, Jeffrey A., M.D.
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: 3 BVT-ASA
Record Dates: First submitted 2010-01-12; First posted 2010-01-13 (Estimated); Last update posted 2015-07-21 (Estimated); Status verified 2015-07

CONDITIONS: Healthy
Keywords: platelet function test; platelets; in vivo test; aspirin; aspirin resistance; aspirin non-responsiveness; in-vivo; To assess the specificity and sensitivity of a novel in-vivo diagnostic test of platelet function; To use this test to define and assess "aspirin resistance"

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patient drinks aspirin in Gatorade. (Active Comparator): Patient drinks Gatorade containing 325 mg aspirin. Bleeding Volume Test is done one hour later.
  Interventions: Drug: Aspirin ingestion followed by doing a Bleeding Volume Test
- Gatorade Placebo (Placebo Comparator): Patient ingests Gatorade and one hour later a Bleeding Volume Test is performed
  Interventions: Procedure: Gatorade Placebo followed by Bleeding Volume Test.

INTERVENTIONS:
Drug: Aspirin ingestion followed by doing a Bleeding Volume Test — Patient drinks a glass of Gatorade containing 325 mg of aspirin, then one hour later a bleeding volume test is performed.
  Arms: Patient drinks aspirin in Gatorade.
Procedure: Gatorade Placebo followed by Bleeding Volume Test. — Patient drinks a glass of Gatorade, then one hour later a bleeding volume test is performed.
  Arms: Gatorade Placebo

SUMMARY:
Purpose of the present research project is to study a new in-vivo test for abnormal platelet function and to study the effect of certain drugs on clinical bleeding. This is a randomized clinical trial of a new in-vivo test of platelet function known as the bleeding volume test(BVT)which relies on an on-line measurement system. This trial will assess the sensitivity and specificity of the new BVT by studying the effects of aspirin which is known to affect platelet function in-vivo. This is not a clinical trial of drugs. This is a clinical trial of a novel in-vivo on-line laboratory test.

The BVT measures the total volume of blood in the discrete blotches of blood on the blotter paper during the BT test and thus the BVT gleans valuable additional information from the bleeding time test (BTT)procedure. We hypothesize that the BV test will be a more accurate, specific and sensitive test for diagnosing platelet function abnormalities and for detecting a person's bleeding tendency compared to the BTT, and commercially available in-vitro platelet function tests.

DETAILED DESCRIPTION:
Purpose of the present research project is to study a new in-vivo test for abnormal platelet function and to study the effect of certain drugs on clinical bleeding. This is a randomized clinical trial of a new in-vivo test of platelet function known as the bleeding volume (BV) test which relies on an on-line measurement system. This trial will assess the sensitivity and specificity of the new BV test by studying the effects of aspirin which is known to affect platelet function in-vivo. This is not a clinical trial of drugs. This is a clinical trial of a novel laboratory test. The BV test results will be compared to the results of two commercially available platelet function tests (the VerifyNow test and the PFA-100 test) which requires 10 ml of blood taken from a peripheral vein.

The bleeding volume test is an extension of the classic Ivy Bleeding Time Test (BTT). The BTT, an in-vivo test for an abnormal bleeding tendency, involves making a small standardized cut in the skin and measuring the duration of bleeding. We hypothesize that measuring both the volume of blood lost (BV) and the BT will to provide a more useful test. The BV test is expected to provide an improved in-vivo technique for 1) investigating the effects of drugs on platelet function and 2) diagnosing diseases of abnormal platelet function such as von Willebrand disease (vWD), 3) identifying patients who are aspirin-resistant in the sense that they do not benefit from the beneficial effects of aspirin in preventing thromboembolic disease (heart attack and stroke), 4) providing insight into the effects of antithrombotic drugs such as clopidogrel, lidocaine and statins (HMG-CoA reductase inhibitors). The BV test will provide an inexpensive diagnostic test and improve patient care.

ELIGIBILITY:
Inclusion Criteria:

* Adult male and female
* Ages 18 to 89 years old

Exclusion Criteria:

* Any history of HIV, Hepatitis C or presence of a blood-borne infectious disease

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2010-01; Primary Completion 2015-10 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Sensitivity, Specificity & ROC curve characteristics of the Bleeding Volume Test | one year

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey A Klein, MD, Principal Investigator — University of Californiia, Riverside
Locations (2):
- United States (2):
  - Private practice office, Newport Beach, California
  - Capistrano Surgery Center, San Juan Capistrano, California